CLINICAL TRIAL: NCT01291368
Title: Does Sedation Influence on Delirium and Post-traumatic Stress-disorder as a Result of Hospitalization in Intensive Care?
Brief Title: Sedation Influence on Delirium and Post-traumatic Stress-disorder as a Result of Hospitalization in Intensive Care
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 1-16-02-50-09
Record Dates: First submitted 2011-01-20; First posted 2011-02-08 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Delirium; Stress Disorders, Post-Traumatic
Keywords: Sedation; Delirium; PTSD; Depression; Anxiety; HRQoL; CAM-ICU; RASS; SF-36; ICU-memory tool; Antipsychotic Agents; Mobilization; ICU-nursing; ICU; intensive care; critical care; critical care nursing
MeSH Terms: conditions — Delirium; Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to investigate if sedation of Intensive Care Unit (ICU) patients influences the development of delirium during their ICU stay and if incidences of delirium have an impact on the development of Post-traumatic Stress-Disorder (PTSD).

Hypothesis 1:

Patients who are minimally sedated, remember staying in ICU and experiences fewer episodes of delirium than patients that are heavily sedated

Hypothesis 2:

Former delirious patients are more likely to develop PTSD

Hypothesis 3:

Delirium decreases health-related quality (HRQoL) of life after discharge

DETAILED DESCRIPTION:
Background:

It is known that ICU patients that experience delirium have longer hospital stay, higher mortality and morbidity. Other studies indicate that PTSD, dementia or depression may emerge after discharge from hospital.

Methods according to hypothesis 1:

During ICU stay: Measure sedation level & delirium. First follow-up 1-2 weeks after ICU: Memories

Analyses:

Data will be analyzed descriptive via EPIDATA and Stata Delirium is endpoint, defined as CAM-ICU positive. Sedation level is exposure variable.

Confounders: priory antipsychotic treatment or hypertension,glasses or hearing aids,alcohol and tobacco abuse,degree of illness,age and sex.

Correlation between sedation level and memories will be calculated.

Methods according to hypothesis 2:

Screening for: PTSD, Depression, Anxiety

Analyses:

PTSD is endpoint, and delirium is the exposure variable. Main confounders: Anxiety and Depression Mean of PTSD will be calculated with Confidence Interval to test any difference between experienced delirium or not.

Methods according to hypothesis 3:

Method:Health-related quality of life is endpoint, Activities of daily living (ADL), Memories, and a Script Test (only after 2 month)

Analyses:

Mean of HRQoL will be calculated with Confidence Interval to test any difference between experienced delirium or not.

Confounders: Diary and/or Follow up

ELIGIBILITY:
Inclusion Criteria:

* ICU-stay > 48 hours

Exclusion Criteria:

* Severe brain trauma
* Non-Danish-speaking
* Age < 18 years
* Death (only hypothesis 2 and 3 in the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients at the ICUs ITA and 600 at Århus Sygehus, Denmark from September 2009 and at Hillerød Intensive, Denmark from 15th October 2010 to 1st October 2011.
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2009-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Sedation level and Delirium | At least twice a day while in the ICU
  Sedation assessed with RASS and delirium assessed with the CAM-ICU by the nurses at the ICU

SECONDARY OUTCOMES:
Post Traumatic Stress Disorder | 2 and 6 month after ICU-discharge
  Minimum 250 patients who accept phone interviews are called twice (after 2 and 6 month) to answer these questionnaires:
  * Intensive Care Unit - memory tool
  * Harvard Trauma Questionnaire (HTQ)
  * Major Depression Inventory (MDI)
  * State-Trait Anxiety Inventory Form Y (STAI)
Health-related quality of life | 2 and 6 month after ICU-discharge
  Minimum 250 patients who accept phone interviews are called twice (after 2 and 6 month) to answer the questionnaires:
  * Activities of daily living (ADL)
  * Short-form 36
  * Script Test (only after 2 month)

CONTACTS AND LOCATIONS:
Overall Officials: Else Tønnesen, MD Professor, Study Chair — Dept. of Anasthesia, Aarhus Universtyhospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Århus Sygehus, Aarhus, Aarhus
  - Anæstesiologisk Afdeling, . Hillerød Hospital, Hillerød, Hillerød